CLINICAL TRIAL: NCT02706808
Title: Effects of Supplementation With Resistant Starch in the Profile of the Intestinal Tract and Cardiovascular Markers in Patients With Chronic Kidney Disease
Brief Title: Resistant Starch Supplementation Effects on the Intestinal Tract Profile and Cardiovascular Markers in Renal Patients
Acronym: Starch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Denise Mafra, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DeniseMafra3
Record Dates: First submitted 2016-02-18; First posted 2016-03-11 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Chronic Kidney Disease; Hemodialysis; Non-dialysis Patients
Keywords: chronic kidney disease; hemodialysis; conservative treatment; resistance starch
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- resistance starch for CKD (Experimental): - Intervention period (6 weeks): Group A - patients will receive 6 cookies/day containing resistant starch (18g/day); Group B - patients will receive 6 cookies/day containing placebo
  Interventions: Dietary Supplement: 'resistance starch for CKD
- cross-over period (Experimental): intervention period (6 weeks): Group B - patients will receive 6 cookies/day containing resistant starch (18g/day); Group A - patients will receive 6 cookies/day containing placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 'resistance starch for CKD — Intervention period (6 weeks): Group A - patients will receive 6 cookies/day containing resistant starch (18g/day); Group B - patients will receive 6 cookies/day containing placebo
  Arms: resistance starch for CKD
Dietary Supplement: Placebo — Intervention period (6 weeks): Group B - patients will receive 6 cookies/day containing resistant starch (18g/day); Group A - patients will receive 6 cookies/day containing placebo
  Arms: cross-over period

SUMMARY:
The objective of this study is to assess whether supplementation with resistant starch from the rice-flour coffee developed by EMBRAPA, as well as from an already industrialized product (Hi-Maize of Ingredion®) could modulate the intestinal microbiota of patients with CKD ( both patients under conservative treatment, such as dialysis treatment), as well as exerting a beneficial effect with respect to reducing levels of inflammatory markers of oxidative stress, uremic toxins and in addition, markers of cardiovascular disease.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD), especially those who are on dialysis have a high prevalence of cardiovascular mortality and, among the risk factors include inflammation and oxidative stress. Recently this scenario, beyond those alterations found in these patients, it has been suggested that the balance of the intestinal flora in these patients might be a new factor of cardiovascular risk. Some treatment strategies have been studied in order to modulate the gut microbiota as the use of pre, pro or synbiotics. Although few studies, supplementation with prebiotics has been recommended. However, the use of resistant starch as a source of prebiotic for modulation of the intestinal flora in these patients has not yet been evaluated, but the study of Prof. Vaziri the University of California Irvine, USA, with nephrectomized rats showed that the resistant starch was able to attenuating the progression of failure of renal function, inflammation and oxidative stress and minimize the abnormalities of intestinal epithelial barrier. The objective of this study is to assess whether supplementation with resistant starch from the rice-flour coffee developed by EMBRAPA, as well as from an already industrialized product (Hi-Maize of Ingredion®) could modulate the intestinal microbiota of patients with CKD ( both patients under conservative treatment, such as dialysis treatment), as well as exerting a beneficial effect with respect to reducing levels of inflammatory markers of oxidative stress, uremic toxins and in addition, markers of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients with arteriovenous fistula as vascular access in the upper limb and on maintenance dialysis for at least 6 months;
* Patients under conservative treatment in stages 3a and 3b (30 to 60 mL / min) of chronic kidney disease and receiving nutritional treatment for at least 6 months (adequate supply of energy 30-35kcal/kg/day and hypoproteic 0.6 g/kg/day.

Exclusion Criteria:

* Patients with autoimmune and infectious diseases, diabetes, cancer and AIDS;
* Patients with catheter for hemodialysis access;
* Patients using catabolizing drugs, supplements as antioxidant vitamin, probiotics, prebiotics, synbiotics and antibiotics.
* Patients who exercise are also deleted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiota profile measured by denaturing gradient gel electrophoresis after supplementation of resistance starch treatment | Change from Baseline microbiota gut at 6 weeks
  after 6 weeks with resistance starch the chronic kidney disease patients should have the gut microbiota modulated
Change in cytokines plasma levels measured by ELISA after supplementation of resistance starch | Change from Baseline inflammation at 6 weeks
  after 6 weeks with resistance starch the chronic kidney disease patients should have the cytokines levels reduced

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, PhD, Principal Investigator — Federal university fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148
- [Derived] Kemp JA, Regis de Paiva B, Fragoso Dos Santos H, Emiliano de Jesus H, Craven H, Z Ijaz U, Alvarenga Borges N, G Shiels P, Mafra D. The Impact of Enriched Resistant Starch Type-2 Cookies on the Gut Microbiome in Hemodialysis Patients: A Randomized Controlled Trial. Mol Nutr Food Res. 2021 Oct;65(19):e2100374. doi: 10.1002/mnfr.202100374. Epub 2021 Aug 22. PMID 34390604